CLINICAL TRIAL: NCT06411392
Title: Stereotactic Antiarrhythmic Radiotherapy for Ventricular Arrhythmia in Austria (Austrian STAR)
Brief Title: SBRT for Ventricular Arrhythmia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35-439 e 22/23
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Ventricular Arrythmia
Keywords: stereotactic radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Antiarrhythmic Radiotherapy (Experimental): Stereotactic antiarrhythmic radiotherapy for refractory ventricular arrhythmia
  Interventions: Radiation: Stereotactic Antiarrhythmic Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Antiarrhythmic Radiotherapy — Patients with ventricular tachycardia will undergo cardiac stereotactic antiarrhythmic radiotherapy with a single fraction of 25 Gy to the arrhythmia substrate, as determined by electrophysiological cardiac mapping.

SUMMARY:
The aim of this study is to demonstrate the safety and efficacy of STAR (Stereotactic Antiarrhythmic Radiotherapy) in patients with VT (ventricular tachycardia) who are unresponsive to standard treatments. Additionally, the planned study aims to provide further insights into the effects of STAR on VT burden, ICD interventions, and insights regarding late toxicities, particularly those related to the heart, which are currently not well understood.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent VTs/VES with significant burden despite guideline-directed therapy
* Existing protective ICD (Implantable cardioverter-defibrillator) implantation except in the presence of contraindications
* AND lack of response or intolerance to antiarrhythmic medication
* AND status post ≥1 catheter ablation due to monomorphic VT(s) and VT early recurrence (<12 months after the last catheter ablation) OR contraindication for endocardial ablation (mechanical valve prosthesis, LV (left ventricular) thrombus, or lack of vascular access in suspicion of endocardial substrate)
* MINIMAL VT BURDEN: The patient must have had at least 3 VT episodes (sustained VT, ICD-ATP, or ICD shock) in the last 3 months prior to study enrollment.
* Presence of suitability for radiation therapy with respect to SBRT
* Age ≥ 18 years
* Existing informed consent

Exclusion Criteria:

* Acute myocardial infarction or percutaneous coronary intervention or heart surgery (<3 months before study enrollment)
* Status post intra-thoracic pre-radiation
* Immediate proximity to radiosensitive structures (e.g., esophagus) making therapy unsafe to administer
* Advanced symptomatic heart failure (NYHA Class IV)
* Polymorphic VT or ventricular fibrillation (confirmed in 12-lead ECG and/or ICD interrogation)
* Extensive myocardial scar substrate that would result in too large of a radiation volume
* Life expectancy < 6 months considering all comorbidities and in the Seattle Heart Failure Model
* Presence of a Left Ventricular Assist Device (LVAD)
* Use of cytotoxic medications
* Pregnancy or lactation - negative pregnancy test within 14 days before study entry required for women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | 30 days
  Demonstration of acute (≤ 30 days) safety of non-invasive stereotactic antiarrhythmic radiotherapy for ventricular arrhythmia (STAR). The primary safety endpoint is defined as ≤ 20% rate of severe adverse events according to CTCAE v5.0 criteria
Efficacy of treatment | 6 months
  The efficacy endpoint is defined by the number of patients experiencing a reduction in ventricular tachycardia episodes, compared to the six-month period prior to SBRT treatment and the six-month period post- SBRT.

SECONDARY OUTCOMES:
Evaluation of changes in the left ventricular ejection fraction | 12 months
  Evaluation of changes in the left ventricular ejection fraction analyzed with echocardiography
Evaluation of mortality | 12 months
  Analysis of cardiac mortality during post-treatment follow-up
Assessment of late side effects | 12 months
  Assessment of radiation-induced cardiac late side effects using late iodine computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volpato G, Compagnucci P, Cipolletta L, Parisi Q, Valeri Y, Carboni L, Giovagnoni A, Dello Russo A, Casella M. Safety and Efficacy of Stereotactic Arrhythmia Radioablation for the Treatment of Ventricular Tachycardia: A Systematic Review. Front Cardiovasc Med. 2022 Aug 22;9:870001. doi: 10.3389/fcvm.2022.870001. eCollection 2022. PMID 36072869
- [Background] Belzile-Dugas E, Eisenberg MJ. Radiation-Induced Cardiovascular Disease: Review of an Underrecognized Pathology. J Am Heart Assoc. 2021 Sep 21;10(18):e021686. doi: 10.1161/JAHA.121.021686. Epub 2021 Sep 6. PMID 34482706
- [Background] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734
- [Background] Loo BW Jr, Soltys SG, Wang L, Lo A, Fahimian BP, Iagaru A, Norton L, Shan X, Gardner E, Fogarty T, Maguire P, Al-Ahmad A, Zei P. Stereotactic ablative radiotherapy for the treatment of refractory cardiac ventricular arrhythmia. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):748-50. doi: 10.1161/CIRCEP.115.002765. No abstract available. PMID 26082532
- [Result] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642